CLINICAL TRIAL: NCT02217800
Title: The Effect of Subcutaneous Infusions of 3 Doses of a Novel Somatostatin Analogue, DG3173, on Growth Hormone Levels in Untreated Acromegalics
Brief Title: The Effect of Subcutaneous Infusions of 3 Doses of DG3173 on Growth Hormone Levels in Untreated Acromegalics
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aspireo Pharmaceuticals Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DG3173-II-02
Record Dates: First submitted 2014-08-14; First posted 2014-08-15 (Estimated); Results first posted 2018-02-15 (Actual); Last update posted 2018-02-15 (Actual); Status verified 2018-01

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly | interventions — Sodium Chloride; PTR 3173; Octreotide

ARMS (1):
- Saline, then DG3173, then octreotide (Other): Interventions: saline, DG3173 and octreotide. Eligible patients are to receive a constant 23 hour subcutaneous infusion of saline as placebo comparator and will be randomized in an equal ratio to one of three treatment sequences of doses of 920, 2760 and 5520 µg DG3173 by constant 23 hour subcutaneous infusions in a random sequence followed by three subcutaneous injections of 300 µg octreotide at approximately 8 hour intervals as an active comparator.
  Interventions: Drug: saline; Drug: DG3173; Drug: octreotide

INTERVENTIONS:
Drug: saline — Eligible patients are to receive a constant 23 hour subcutaneous infusion of saline as placebo comparator and will be randomized in an equal ratio to one of three treatment sequences of doses of 920, 2760 and 5520 µg DG3173 by constant 23 hour subcutaneous infusions in a random sequence followed by three subcutaneous injections of 300 µg octreotide at approximately 8 hour intervals as an active comparator.
Drug: DG3173 — Eligible patients are to receive a constant 23 hour subcutaneous infusion of saline as placebo comparator and will be randomized in an equal ratio to one of three treatment sequences of doses of 920, 2760 and 5520 µg DG3173 by constant 23 hour subcutaneous infusions in a random sequence followed by three subcutaneous injections of 300 µg octreotide at approximately 8 hour intervals as an active comparator.
Drug: octreotide — Eligible patients are to receive a constant 23 hour subcutaneous infusion of saline as placebo comparator and will be randomized in an equal ratio to one of three treatment sequences of doses of 920, 2760 and 5520 µg DG3173 by constant 23 hour subcutaneous infusions in a random sequence followed by three subcutaneous injections of 300 µg octreotide at approximately 8 hour intervals as an active comparator.

SUMMARY:
This study is designed to assess the effect of the different continuous s.c. infusion treatments on the human growth hormone (hGH) levels in untreated acromegalic patients in comparison to a standard dose of octreotide. In addition, the pharmacokinetic profile and the safety and tolerability of DG3173 after continuous s.c. infusion will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Men, women of non child-bearing potential, or women of child-bearing potential who either abstain from sexual intercourse, have a sterile partner or practice two medically approved, non-hormonal methods of contraception
* Diagnosis of acromegaly of pituitary origin
* Have an age-adjusted insulin-like growth factor type 1 (IGF-1) concentration ≥1.2 times the upper limit of normal range on at least one measurement in the 12 months prior to screening (Visit 1) AND a second raised value screening
* Have at least one random hGH level of ≥5 μg/L in the 12 months prior to screening AND a second raised value at screening
* Have given written informed consent
* Ability to comply with the requirements of the protocol for the study

Exclusion Criteria:

* Previous specific treatment for acromegaly in the 12 months prior to screening, including somatostatin analogues (SSAs); surgery; radiotherapy and pegvisomant
* Treatment with dopamine agonists in the 3 months prior to screening
* Uncontrolled hypertension
* Type I diabetes mellitus, poorly-controlled type II diabetes mellitus (glycosylated haemoglobin [HbA1c] ≥7.5%) and patients requiring insulin treatment
* Gallstones or gravel that could cause biliary obstruction
* Hyperprolactinaemia
* Participation in a clinical study within 60 days prior to screening
* Receipt of blood, blood products or plasma derivatives 60 days prior to screening
* Body mass index (BMI) below 22 or above 37 kg/m2
* Pregnancy, lactation or use of any hormonal based contraceptives
* Concomitant intake of corticosteroids or levodopa
* A history of active alcohol abuse or drug addiction
* Positive viral serology screening result for hepatitis B surface antigen, antibodies to hepatitis C virus, or human immunodeficiency virus type 1 and 2
* Evidence or suspicion of tumour expansion
* Clinically significant abnormality in screening ECG in the opinion of the Investigator
* Any clinically significant abnormal in screening laboratory safety test (biochemistry, haematology and dipstick urinalysis) in the opinion of the Investigator
* Any disease which in the Investigator's opinion would exclude the patient from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-11; Primary Completion 2014-03 (Actual); Study Completion 2016-05 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Saline, Then DG3173, Then Octreotide
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Saline, Then DG3173, Then Octreotide
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3
Region of Enrollment [Number; unit: participants]
  Ukraine | 8

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients Who Achieve a Trough Human Growth Hormone (hGH) Concentration of <2.5µg/L During the Last 12 Hours of the 23 Hour Profile Following Each Study Treatment.
Time Frame: 23 hours following each treatment
Measure: Number; unit: participants with trough hGH < 2.5 µg/mL
Arm/Group | Saline (Control) | 920 µg DG3173 | 2760 µg DG3173 | 5520 µg DG3173 | Active Control (Octreotide)
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
participants with trough hGH < 2.5 µg/mL | 0 | 1 | 2 | 3 | 4

ADVERSE EVENTS:
Arm/Group | Saline (Control) | 920 µg DG3173 | 2760 µg DG3173 | 5520 µg DG3173 | Active Control (Octreotide)
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 1/8 | 1/8 | 2/8 | 2/8 | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Saline (Control) (N=8) | 920 µg DG3173 (N=8) | 2760 µg DG3173 (N=8) | 5520 µg DG3173 (N=8) | Active Control (Octreotide) (N=8)
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 1 | 2 | 2 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No